CLINICAL TRIAL: NCT04274517
Title: The Effect of Dilute Chlorhexidine Versus Betadine on Microbial Growth in Operative Splash Basins During Total Joint Arthroplasty: A Prospective Clinical Trial
Brief Title: Microbial Growth in Operative Splash Basins During Total Joint Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary analysis showed lack of positive finding, indicating a substantial number of subjects required, which is not feasible based on budget and timeline.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Nathanael Heckmann, Assistant Professor of Clinical Orthopaedic Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS-19-01005
Record Dates: First submitted 2020-02-12; First posted 2020-02-18 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Periprosthetic Joint Infection
MeSH Terms: interventions — Povidone-Iodine; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know which treatment arm they have been randomized to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Sterile Water (Experimental)
  Interventions: Other: Sterile Water
- 3.5% betadine (Experimental)
  Interventions: Other: 3.5% Betadine
- 0.05% chlorhexidine gluconate (Experimental)
  Interventions: Other: 0.05% Chlorhexidine Gluconate

INTERVENTIONS:
Other: Sterile Water — 1L of sterile water used in surgical splash basins during total joint arthroplasty to clean surgical instrumentation.
  Arms: Sterile Water
Other: 3.5% Betadine — 1L of 3.5% betadine used in surgical splash basins during total joint arthroplasty to clean surgical instrumentation.
  Arms: 3.5% betadine
Other: 0.05% Chlorhexidine Gluconate — 1L of clorhexidine gluconate used in surgical splash basins during total joint arthroplasty to clean surgical instrumentation.
  Arms: 0.05% chlorhexidine gluconate

SUMMARY:
The usage of splash basins in the setting of total knee arthroplasty and total hip arthroplasty presents a risk of contamination and subsequent periprosthetic joint infection. Previous studies have investigated the efficacy of multiple antimicrobial irrigants for preventing periprosthetic joint infection, but the results are varied.

Despite several noteworthy studies on the appropriate usage of different antiseptic solutions in surgical splash basins, the current literature has several limitations. First, there are no head-to-head clinical trials comparing betadine and chlorhexidine gluconate (CHG) usage with relation to periprosthetic joint infection and splash basin contamination rates. Second, the in vitro studies directly cultured splash basin antiseptic solutions rather than culturing surgical instruments.

The objective of this study is to compare the microbial contamination rate of total joint arthroplasty instruments that have been placed in surgical splash basins filled with either sterile water, 3.5% betadine, or 0.05% CHG. The overall purpose of the study is to investigate the efficacy of 0.05% CHG and determine if it is an appropriate solution to use in surgical splash basins for joint replacement surgeries.

A prospective clinical trial will be conducted. Patients treated at the Keck Hospital of USC or USC Verdugo Hills Hospital for primary total hip or total knee arthroplasty will be screened for inclusion in our study. All primary surgeries will be performed according to the preferences of the operating surgeon. No deviations from standard surgical care will be made based on inclusion in this study. However, prior to surgery, patients who elect to participate will be randomized to one of three groups: (1) sterile water, (2) 3.5% betadine, or (3) 0.05% CHG.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to Keck Hospital of USC or USC Verdugo Hills Hospital for primary total knee arthroplasty or total hip arthroplasty.

Exclusion Criteria:

* Age < 18 years.
* History of previous total hip arthroplasty or total knee arthroplasty.
* History of previous knee or hip joint infection.
* History of previous allergic reaction to chlorhexidine.
* Known allergy to iodine or shellfish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Microbial Contamination Rate of Surgical Instruments | 14 days
  Microbial contamination rate of total joint arthroplasty instruments that have been placed in surgical splash basins filled with either sterile water, 3.5% betadine, or 0.05% CHG

SECONDARY OUTCOMES:
90-Day Wound Complication | 90 days
  Differences in 90-day wound complications and 90-day periprosthetic joint infections between the sterile water, 3.5% betadine, and 0.05% CHG surgical splash basin groups

CONTACTS AND LOCATIONS:
Locations (1):
- Keck School of Medicine of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anto B, McCabe J, Kelly S, Morris S, Rynn L, Corbett-Feeney G. Splash basin bacterial contamination during elective arthroplasty. J Infect. 2006 Mar;52(3):231-2. doi: 10.1016/j.jinf.2005.06.013. Epub 2005 Dec 28. No abstract available. PMID 16386799
- [Background] Baird RA, Nickel FR, Thrupp LD, Rucker S, Hawkins B. Splash basin contamination in orthopaedic surgery. Clin Orthop Relat Res. 1984 Jul-Aug;(187):129-33. PMID 6744706
- [Background] Frisch NB, Kadri OM, Tenbrunsel T, Abdul-Hak A, Qatu M, Davis JJ. Intraoperative chlorhexidine irrigation to prevent infection in total hip and knee arthroplasty. Arthroplast Today. 2017 May 12;3(4):294-297. doi: 10.1016/j.artd.2017.03.005. eCollection 2017 Dec. PMID 29204500